CLINICAL TRIAL: NCT05344950
Title: Development and Pilot Testing of AURA
Brief Title: Connecting Audio and Radio Sensing Systems to Improve Care at Home
Acronym: AURA
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency); National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC2123
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Bladder Cancer; Ovarian Cancer; Cervical Cancer; Uterine Cancer
Keywords: ostomy (colostomy, urostomy, and ileostomy); symptom; self-management; caregiving; family research; telehealth; self-efficacy; quality of life; post-treatment care transition
MeSH Terms: conditions — Colorectal Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — Radio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AURA: In addition to usual care, participants assigned to this arm will have access to our Audio + Radio (AURA) system.
  Interventions: Behavioral: Audio + Radio (AURA)

INTERVENTIONS:
Behavioral: Audio + Radio (AURA) — Participants will receive personalized self-care information based on their symptoms and signs of complications (e.g., fatigue) from interacting with our voice assistant device, connected to a system that integrating the patient-reported outcome and objective data from passive RF sensing to provide continuous monitoring of patients' symptoms and complications after they are discharged home.

SUMMARY:
This study aims to assess the usability of the innovative Audio + Radio (AURA) system in enhancing personalized supportive care for cancer patients and caregivers during the post-ostomy care transition by collecting information on patient's daily activities and answers to survey questionnaire, and enabling access to this information through a voice assistant device.

DETAILED DESCRIPTION:
The investigators will assign up to 30 cancer patients with newly created ostomies for cancer treatment with curative intent and their primary caregivers to the AURA or usual care groups (up to 30 patient-caregiver dyads, a total of 60 individuals). AURA is defined as a system that connects audio-based voice assistant devices with radiofrequency (RF) sensing technology to gather relevant patient information automatically, interactively, and with context-awareness and to store a patient's health records that otherwise had to be measured and entered manually into an electronic system. Additionally, the system enables user's access to this information through a voice assistant device. The users of this system will be the entire care team, consisting of the patient and their family members as well as the caregivers and healthcare providers at remote sites. If results indicate that the pilot trial is feasible, the investigators will design and conduct a definitive trial to examine the efficacy of AURA, a potentially scalable intervention that can be disseminated through oncology clinics nationwide to enhance post-treatment care for cancer patients with ostomies who transition from hospital professional care to self-management at home and their caregivers.

ELIGIBILITY:
Inclusion Criteria

Phase I: The investigators will only be recruiting patients for this phase

Patients must:

* have been surgically treated for colorectal or bladder cancer with curative intent;
* have had an ostomy with curative intent for at least 90 days;
* be able to read and speak English;
* be 18 years or older;

Phase II: The investigators will be recruiting patients and caregivers as a dyad for this phase

* Patients must:

  * have been surgically treated for colorectal or bladder cancer with curative intent;
  * be within one month of hospital discharge of a newly created ostomy with curative intent;
  * be able to read and speak English;
  * be 18 years or older;
  * have a caregiver who is willing to participate in the study;
* Caregivers must:

  * be 18 years or older;
  * be able to read and speak English;
  * be identified as the primary caregiver by the patient;
  * have not themselves been diagnosed with cancer or received cancer treatment during the study (to ensure that patients and caregivers focus their efforts on care of the patient).

Exclusion Criteria

Patients and their caregivers will be excluded if they:

* are unable to read, speak, or understand English;
* have more than one type of ostomy;
* have other cancer diagnosis (excluding non-melanomatous skin cancer); or
* have cognitive impairment (assessed by the Short Portable Mental Status Questionnaire).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects receive treatment and their caregivers partners.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the AURA system | 1-month followup survey
  Satisfaction with the AURA system will be assessed by the 9-item Participant Satisfaction Scale measuring the level of program satisfaction ranging from 1=not satisfied to 5=extremely satisfied. Higher total score indicates greater program satisfaction.
Perceived ease of use of the PRISMS program | 1-month followup survey
  Perceived ease of use of the AURA system will be assessed by the 23-item Usability Scale measuring the ease of use in three aspects: general, content, and navigation. The scales range from 1=strongly disagree to 5=strongly agree. Higher total score indicates greater ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Shahriar Nirjon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UT Health San Antonio MD Anderson Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
This is a pilot study with very small sample size and specific inclusion criteria. Sharing data with others may increase the risk to patient confidentiality.

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials